CLINICAL TRIAL: NCT03856866
Title: Hydroxychloroquine Administration for Reduction of Pexophagy
Acronym: HARP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Neal Sondheimer, Staff Physician - Clinical and Metabolic Genetics, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1000061385
Record Dates: First submitted 2018-11-05; First posted 2019-02-27 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Zellweger Syndrome; Peroxisome Biogenesis Disorders
Keywords: PBD, Zellweger spectrum, PBD-ZSD
MeSH Terms: conditions — Zellweger Syndrome; Peroxisome biogenesis disorders | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: A randomized, blinded, placebo controlled, crossover N of 1 trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties will be masked except for research pharmacy who will do the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hydroxychloroquine (Experimental): Hydroxychloroquine: liquid suspension, 4mg/kg/day by mouth, divided bid for 84 days.
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Liquid suspension compounded to mimic the taste, appearance and texture of the investigational agent.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine: 4mg/kg/day, divided bid.
  Other Names: Apo-Hydroxyquine; Plaquenil
  Arms: Hydroxychloroquine
Drug: Placebo — Liquid suspension compounded to mimic the active hydroxycholoquine interventional agent.
  Arms: Placebo

SUMMARY:
A series of N-of-1, crossover, randomized, placebo-controlled, double-blinded trial. Hydroxychloroquine (HCQ) and a crossover to placebo (order is randomized and blinded) will be administered in liquid suspension for 84 days (12 weeks) each with an 84 day washout in between. We hypothesize that HCQ will reduce peroxisomal turnover, which will arrest ongoing injury in PBDs caused by PEX1, PEX6 or PEX26.

DETAILED DESCRIPTION:
HARP is a phase II/III, double-blind, placebo-controlled, randomized, crossover series N-of-1 study of the effect of hydroxychloroquine (HCQ) in patients with peroxisomal biogenesis disorders (PBD-ZSD). Patients eligible for the study must have a laboratory diagnosis of PEX1, PEX6 or PEX26 dependent PBD-ZSD from a CLIA or SCC-certified clinical laboratory, a history of abnormal VLCFA levels, and must be at least 84 days from their last HCQ dose. Patients will be excluded for known sensitivity to HCQ, known glucose-6-phosphate dehydrogenase deficiency, if they have an expected survival of less than 9 months or if they are participating in another interventional clinical trial.

HCQ will be administered at a dose of 4mg/kg/day divided into two doses, as a liquid suspension that can be given orally or through nasogastric or gastric tube. Within the study, HCQ or placebo will be given for 84 days, followed by a washout period of 84 days followed by an 84 day crossover to the alternative therapy to assess the effect the study measures.

Study measures will be completed at four intervals (initiation, end of period 1, start of period 2, end of trial). Ophthalmological monitoring of patients has three components, electroretinogram (ERG), visual acuity testing and optical coherence tomography (OCT). Plasma levels of very long-chain fatty acids (VLCFA), plasmalogen and phytanic acid will be assessed. Parents will also be administered The Pediatric Inventory for Parents (PIP), a questionnaire that was developed to evaluate the stress associated with parenting a seriously ill child, at the end of period 1 and period 2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a peroxisomal defect due to PEX1, PEX6 or PEX26 through a SCC or CLIA-certified clinical genetic testing laboratory.
* Abnormal plasma very-long-chain fatty acid levels.
* All therapies available in Canada have been considered and ruled out, have failed or were justified as being unsuitable for the patient. We note that there are no therapies available.
* At least 84 days from last HCQ dose

Exclusion Criteria:

* Known sensitivity to HCQ.
* Known Glucose-6-phosphate dehydrogenase deficiency.
* Expected survival is less than six months.
* The patient does not provide informed consent.
* The patient is participating in another interventional clinical trial.

Ages: 6 Months to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Electroretinogram (ERG) voltage changes. | 12 week. Measurements at Day 0, Day 84(+/-7 days) of each treatment arm.
  Electroretinograms are a diagnostic test that measures the electric activity within cells in response to stimulus. ERG voltages are depressed in peroxisomal disease, and the quantitative evaluation of ERG voltage is another measure that has been used as an endpoint for clinical trials in peroxisomal disease. Change in b-wave voltage before and after treatment period.
Change in the red blood cell levels of plasmalogen. | 12 week. Measurements at Day 0, Day 84(+/-7 days) of each treatment arm.
  Change in the red blood cell levels of plasmalogen (18:0 dimethylacetals/18:0 ratio).
Change in the plasma levels of phytanic acid. | 12 week. Measurements at Day 0, Day 84(+/-7 days) of each treatment arm.
  Change in the plasma levels of phytanic acid.
Change in the plasma levels of very-long chain fatty acids. | 12 week. Measurements at Day 0, Day 84(+/-7 days) of each treatment arm.
  Change in the plasma levels of very-long chain fatty acids (C26/C22).

SECONDARY OUTCOMES:
Eye examination: Optical Coherence Tomography | 12 week. Measurements at Day 0, Day 84(+/-7 days) of each treatment arm.
  Optical coherence tomography is an imaging study of the retina. OCT is routinely performed in clinical management of patients with peroxisomal disease.
Eye examination: Visual Acuity | 12 week. Measurements at Day 0, Day 84(+/-7 days) of each treatment arm.
  Visual acuity testing evaluates the visual performance of patients using the reading of a logMAR chart. Visual acuity testing is routinely performed in clinical management of patients with peroxisomal disease.
Pediatric Inventory for Parents (PIP) following the treatment arms. | 36 week. Measurements following each treatment arm.
  The PIP is a validated measure of parental stress related to the care for children with chronic illness.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Sondheimer, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided